CLINICAL TRIAL: NCT02179008
Title: Multi-center Phase II Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension
Acronym: SEE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33-003
Record Dates: First submitted 2014-06-26; First posted 2014-07-01 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Santen; Eye; Glaucoma; Ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- DE-117 Low Dose ophthalmic solution (Experimental): One drop Low Dose DE-117 in each eye QD for 90 days
  Interventions: Drug: DE-117 Low Dose ophthalmic solution
- DE-117 Low/Middle Dose ophthalmic solution (Experimental): One drop DE-117 Low/Middle Dose ophthalmic solution in each eye QD for 90 days
  Interventions: Drug: DE-117 Low/Middle Dose ophthalmic solution
- DE-117 Middle Dose ophthalmic solution (Experimental): One drop Middle Dose DE-117 in each eye QD for 90 days
  Interventions: Drug: DE-117 Middle Dose ophthalmic solution
- DE-117 Middle/High Dose ophthalmic solution (Experimental): One drop Middle/High Dose DE-117 in each eye QD for 90 days
  Interventions: Drug: DE-117 Middle/High Dose ophthalmic solution
- DE-117 High Dose ophthalmic solution (Experimental): One drop High Dose DE-117 in each eye QD for 90 days
  Interventions: Drug: DE-117 High Dose ophthalmic solution
- latanoprost ophthalmic solution 0.005% (Active Comparator): One drop latanaprost in each eye QD for 90 days
  Interventions: Drug: latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: DE-117 Low Dose ophthalmic solution — Low Dose DE-117 ophthalmic solution
  Other Names: DE-117
  Arms: DE-117 Low Dose ophthalmic solution
Drug: DE-117 Low/Middle Dose ophthalmic solution — Low/Middle Dose DE-117
  Other Names: DE-117
  Arms: DE-117 Low/Middle Dose ophthalmic solution
Drug: DE-117 Middle Dose ophthalmic solution — Middle Dose DE-117
  Other Names: DE-117
  Arms: DE-117 Middle Dose ophthalmic solution
Drug: DE-117 Middle/High Dose ophthalmic solution — Middle/High Dose DE-117
  Other Names: DE-117
  Arms: DE-117 Middle/High Dose ophthalmic solution
Drug: DE-117 High Dose ophthalmic solution — High Dose DE-117
  Other Names: DE-117
  Arms: DE-117 High Dose ophthalmic solution
Drug: latanoprost ophthalmic solution 0.005% — 0.005% latanoprost
  Other Names: latanoprost
  Arms: latanoprost ophthalmic solution 0.005%

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of five concentrations of DE-117 ophthalmic solution.

DETAILED DESCRIPTION:
This is a 90-day randomized, observer-masked, active-controlled, parallel-group, multi-center, study assessing the safety and efficacy of five concentrations of DE-117 ophthalmic solution when compared to latanoprost (0.005% latanoprost) in subjects with primary open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of primary open-angle glaucoma or ocular hypertension in both eyes
* Qualifying intraocular pressure in at least one eye at Baseline
* Qualifying corrected ETDRS visual acuity in each eye
* Qualifying central cornea thickness in each eye

Exclusion Criteria:

* Closed/barely open anterior chamber angle or a history of acute angle closure in either eye
* Diagnosis of primary open-angle glaucoma or ocular hypertension due to etiology known to be non-responsive to conventional drug therapy
* Evidence of advanced glaucoma, visual field defect or progressive visual field loss that that do not meet the study criteria
* History of ocular surgery specifically intended to lower IOP
* History of any ocular or systemic abnormality or condition that may put the subject at significant risk, may confound study results, or may interfere significantly with the subject's participation in the study
* Intended or current use of any ocular medications other than study medications during the study
* Use of contact lenses within one week prior to Baseline (Day 1) until end of treatment
* Known allergy or sensitivity to any components of the study medications
* Use of steroids (systemic) within 30 days prior to Visit 1 (Screening)
* Anticipate the need to initiate or modify an existing chronic therapy that could substantially affect IOP or the study outcomes during the study period
* Females who are pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (mmHg) | Day 91
  Intraocular pressure (mmHg) measurements will be collected using Goldmann applanation tonometry

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as a Measure of Safety and Tolerability | Day 1, Day 8, Day 15, Day 31, Day 61 and Day 91
  Adverse events will be assessed at each visit to evaluate safety

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Chandler, Arizona
  - Artesia, California
  - Glendale, California
  - Long Beach, California
  - Newport Beach, California
  - Largo, Florida
  - Morrow, Georgia
  - Roswell, Georgia
  - Rochester, New York
  - High Point, North Carolina
  - Cleveland, Ohio
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas